CLINICAL TRIAL: NCT04563442
Title: Comorbidities And Complications Associated With Covid-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Gamal Hussein, Principal investigator, Assiut University
Other Study IDs: covid 19
Record Dates: First submitted 2020-09-23; First posted 2020-09-24 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- covid 19: complications and comorbidities
  Interventions: Other: complication

INTERVENTIONS:
Other: complication — complication co morbidities

SUMMARY:
To evaluate the spectrum of comorbidities and complications and its impact on the clinical outcome in hospitalized patients with coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
Severe acute respiratory syndrome (SARS) coronavirus 2 (SARS-CoV-2) is a coronavirus with human infection designated as COVID-19 by the World Health Organization. Bats and birds serve as the typical coronavirus hosts, with zoonotic spread and a long-documented history of animal-animal-human transmission.

Since November 2019, the rapid outbreak of coronavirus disease 2019 (COVID-19), which arose from severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, has recently become a public health emergency of international concern. COVID-19 has contributed to an enormous adverse impact globally.

As of 10 March 2020 there have been 113702 laboratory confirmed cases and 4012 deaths globally.

According to the latest reports, the clinical manifestations of COVID-19 are heterogeneous. On admission, 20-51% of patients were reported as having at least one comorbidity, with diabetes (10-20%), hypertension (10-15%) and other cardiovascular and cerebrovascular diseases (7-40%) being most common. Previous studies have demonstrated that the presence of any comorbidity has been associated with a 3.4-fold increased risk of developing acute respiratory distress syndrome in patients with H7N9 infection. As with influenza, SARS-CoV and Middle East Respiratory Syndrome coronavirus (MERS-CoV), COVID-19 is more readily predisposed to respiratory failure and death in susceptible patients.

Although it is well documented that COVID-19 is primarily manifested as a respiratory tract infection, emerging data indicate that it should be regarded as a systemic disease involving multiple systems, including cardiovascular, respiratory, gastrointestinal, neurological, hematopoietic and immune system. Mortality rates of COVID-19 are lower than SARS and Middle East Respiratory Syndrome (MERS); however, COVID-19 is more lethal than seasonal flu.

Older people and those with comorbidities are at increased risk of death from COVID-19, but younger people without major underlying diseases may also present with potentially lethal complications such as fulminant myocarditis and disseminated intravascular coagulopathy (DIC).

ELIGIBILITY:
Inclusion Criteria:

Patients presented by respiratory symptom and admitted to Assuit university hospitals in wards and intensive care units due to COVID-19 according to WHO and Egyptian Ministry of Health and Population (MOH) definitions with positive PCR result.

Exclusion Criteria:

* Negative PCR result for suspicious cases of Covid-19,
* Patients refusing to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients confirmed to have covid 19 infection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-25 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-02-25 (Estimated)

PRIMARY OUTCOMES:
Effect of different comorbidities and covid-19 infection' complications on patient's outcome | baseline
  Identifying characters of patients with covid-19 whose are susceptible to have different complications during the course of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Mohamed Rabee, Proffessor, Study Chair — Assuit university hospital

REFERENCES:
- [Result] Layton DS, Choudhary A, Bean AGD. Breaking the chain of zoonoses through biosecurity in livestock. Vaccine. 2017 Oct 20;35(44):5967-5973. doi: 10.1016/j.vaccine.2017.07.110. Epub 2017 Aug 18. PMID 28826750
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Gao HN, Lu HZ, Cao B, Du B, Shang H, Gan JH, Lu SH, Yang YD, Fang Q, Shen YZ, Xi XM, Gu Q, Zhou XM, Qu HP, Yan Z, Li FM, Zhao W, Gao ZC, Wang GF, Ruan LX, Wang WH, Ye J, Cao HF, Li XW, Zhang WH, Fang XC, He J, Liang WF, Xie J, Zeng M, Wu XZ, Li J, Xia Q, Jin ZC, Chen Q, Tang C, Zhang ZY, Hou BM, Feng ZX, Sheng JF, Zhong NS, Li LJ. Clinical findings in 111 cases of influenza A (H7N9) virus infection. N Engl J Med. 2013 Jun 13;368(24):2277-85. doi: 10.1056/NEJMoa1305584. Epub 2013 May 22. PMID 23697469
- [Result] Placzek HE, Madoff LC. Association of age and comorbidity on 2009 influenza A pandemic H1N1-related intensive care unit stay in Massachusetts. Am J Public Health. 2014 Nov;104(11):e118-25. doi: 10.2105/AJPH.2014.302197. Epub 2014 Sep 11. PMID 25211746
- [Result] Mauskopf J, Klesse M, Lee S, Herrera-Taracena G. The burden of influenza complications in different high-risk groups: a targeted literature review. J Med Econ. 2013;16(2):264-77. doi: 10.3111/13696998.2012.752376. Epub 2012 Dec 4. PMID 23173567
- [Result] Booth CM, Matukas LM, Tomlinson GA, Rachlis AR, Rose DB, Dwosh HA, Walmsley SL, Mazzulli T, Avendano M, Derkach P, Ephtimios IE, Kitai I, Mederski BD, Shadowitz SB, Gold WL, Hawryluck LA, Rea E, Chenkin JS, Cescon DW, Poutanen SM, Detsky AS. Clinical features and short-term outcomes of 144 patients with SARS in the greater Toronto area. JAMA. 2003 Jun 4;289(21):2801-9. doi: 10.1001/jama.289.21.JOC30885. Epub 2003 May 6. PMID 12734147
- [Result] Driggin E, Madhavan MV, Bikdeli B, Chuich T, Laracy J, Biondi-Zoccai G, Brown TS, Der Nigoghossian C, Zidar DA, Haythe J, Brodie D, Beckman JA, Kirtane AJ, Stone GW, Krumholz HM, Parikh SA. Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the COVID-19 Pandemic. J Am Coll Cardiol. 2020 May 12;75(18):2352-2371. doi: 10.1016/j.jacc.2020.03.031. Epub 2020 Mar 19. PMID 32201335